CLINICAL TRIAL: NCT00077727
Title: A Study of Galantamine HBr as an Adjunctive Treatment to Atypical Antipsychotic Medications in Outpatients With Schizophrenia and Associated Cognitive Deficits.
Brief Title: A Study of the Effectiveness and Safety of Galantamine Hydrobromide on Cognitive Impairment in Patients With Schizophrenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR004366
Record Dates: First submitted 2004-02-11; First posted 2004-02-16 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; cognitive impairment; galantamine; acetylcholinesterase inhibitors; antipsychotic drugs; BACS
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

INTERVENTIONS:
Drug: Extended-release galantamine hydrobromide

SUMMARY:
The purpose of this study is to determine if adding extended-release galantamine hydrobromide, compared with adding placebo, to current atypical antipsychotic therapy is well tolerated and effective in improving cognitive impairment in patients with schizophrenia.

DETAILED DESCRIPTION:
Galantamine acts on acetylcholinesterase, and has been shown to effectively treat cognitive symptoms in patients with Alzheimer's disease. Previous cellular research of nicotinic receptors has shown promising results, and it is theorized that the nicotinic system of patients with schizophrenia may be abnormal and may play an important role in the cognitive symptoms associated with schizophrenia. It is also postulated that galantamine may improve neuropsychiatric symptoms such as hallucinations, delusions, and apathy in patients with Alzheimer's disease. Atypical antipsychotic medications are effective treatment for schizophrenia patients but some symptoms remain. Therefore, galantamine may be a useful cotreatment for schizophrenia patients on atypical antipsychotic treatment. This is a pilot dose-ranging, randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), placebo-controlled multicenter study that examines the effects of taking extended-release galantamine hydrobromide (16 or 24 mg once daily) or placebo on the effectiveness in reducing symptoms of schizophrenia patients who are already taking an atypical antipsychotic medication. The safety of combined treatment is also examined. Measures of effectiveness include the Positive and Negative Syndrome Scale (PANSS) to measure neuropsychiatric symptoms of schizophrenia; the Clinical Global Impression (CGI) scale to measure change over the course of the study; the Brief Assessment of Cognition in Schizophrenia (BACS) for verbal memory and learning, working memory, motor function, attention, verbal fluency, and executive functioning; the Continuous Performance Test (CPT) for sustained attention and distractability; reaction time test (RTT) and finger tapping test (FTT) for psychomotor speed; Lexical and Semantic Fluency Test (LSFT) for language skills. As schizophrenia patients are a population with high nicotine use, and galantamine may act on nicotine receptors, blood levels of nicotine are also measured as varying nicotine levels could alter the effects of galantamine. The null hypothesis that there is no difference between the 2 groups (galantamine cotreatment and placebo) will be tested for each of the efficacy measurements (total PANSS, BACS, and CGI scores) at Week 8. Measures of safety include physical examinations, electrocardiograms (ECGs), clinical laboratory tests, measurement of plasma prolactin concentrations, pregnancy test for women, and incidence of adverse events. Adverse events that might be related to the medications are also monitored using the Simpson-Angus Extrapyramidal Side Effects Scale (SAS), the Barnes Akathisia Rating Scale (BARS), and the Abnormal Involuntary Movement Scale (AIMS). Extended-release galantamine hydrobromide or matching placebo capsules for once-daily dosing. Patients take 8 milligrams (mg) per day during Week 1, 16 mg per day during Week 2, and 16 mg or 24 mg per day (depending on randomization) during Weeks 3 to 8. Treatment groups are placebo capsule, 16 mg capsule, 24 mg capsule.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia present for at least 1 year, and has not returned to his/her level of functioning before the disease, with a Brief Psychiatric Rating Scale score of 30 to 60 (inclusive), and cognitive impairment as determined by scores from neuropsychological tests and subtests
* Nicotine user with a minimum intake equivalent to 5 cigarettes per day
* On a stable dose of allowed atypical antipsychotic medication (risperidone [either oral or CONSTA], olanzapine, quetiapine, ziprasidone, or aripiprazole) alone or in combination, for at least 30 days before screening, and deemed able to continue on the same dose
* Women patients must be postmenopausal, surgically sterile, or using appropriate contraception before entry and throughout the study, and have a negative pregnancy test at screening
* Able to read, write, and understand English, and has no limitations in communication skills that would prevent him/her from completing the cognitive tests used in this study.

Exclusion Criteria:

* Previously enrolled in a galantamine hydrobromide study
* Any clinically significant uncontrolled medical illness (such as peptic ulcer disease
* urinary tract obstruction
* or neurologic, cardiac, hepatic, renal, metabolic, or endocrine disturbances)
* History of severe asthma
* Any history of epilepsy or convulsions, except for febrile convulsions during childhood
* History of cancer within the past year, except for treated basal cell carcinoma, or any history of prolactin-dependent breast cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2003-03; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The key exploratory efficacy end points are the change from baseline to Week 8 in total PANSS score, total BACS score, and CGI global improvement and severity of illness scores.

SECONDARY OUTCOMES:
Additional efficacy assessments included subscore analyses for LSFT, CPT, RTT and FTT.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the effectiveness and safety of galantamine hydrobromide on cognitive impairment in patients with schizophrenia. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1085&filename=CR004366_CSR.pdf